CLINICAL TRIAL: NCT02015221
Title: Evaluation of a Dual Action Pneumatic Compression Device: Patient Ease of Use and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tactile Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ACTitouch EOU
Record Dates: First submitted 2013-12-02; First posted 2013-12-19 (Estimated); Results first posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Venous Insufficiency
Keywords: chronic venous insufficiency; venous leg ulcers; pneumatic compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACTitouch (Experimental): ACTitouch in sustained gradient compression mode during all waking hours (at least 10 hours per day) and intermittent pneumatic compression mode for 2 hours each day.
  Interventions: Device: Dual Action Pneumatic Compression Device
- Standard Compression Garments (Active Comparator): Standard Compression Garments of compression levels 30mmHg to 40mmHg during all waking hours each day.
  Interventions: Device: Standard Compression Garments

INTERVENTIONS:
Device: Dual Action Pneumatic Compression Device — A novel dual action pneumatic compression device that provides both sustained compression while ambulatory, and intermittent pneumatic compression when connected to an AC outlet.
  Arms: ACTitouch
Device: Standard Compression Garments — Compression stockings with a 30-40mmHg level of compression.
  Arms: Standard Compression Garments

SUMMARY:
The purpose of this study is to determine the ease of use and comfort of the ACTitouch dual action pneumatic compression device in patients with unilateral or bilateral chronic venous insufficiency (CVI) with or without venous leg ulcers, as compared to standard compression.

DETAILED DESCRIPTION:
Subjects will be randomized to receive either the ACTitouch system or standard compression garments, and will respond to symptom surveys and quality of life surveys to assess comfort and ease of use of each. These will be conducted at Baseline, at Day 15 and Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral or bilateral CVI with or without leg ulcers
* Documented history of low adherence to compression garment therapy
* CEAP classification C3-C6
* Leg circumferences within the following ranges: Ankle 12-44cm, calf 22-6m, below the knee 22-68cm

Exclusion Criteria:

* History of skin sensitivity to any of the components of ACTitouch or compression garments
* History of acute (deep vein thrombosis) DVT or (pulmonary embolism) PE within the last 3 months
* Ankle Brachial Index (ABI) < 0.8
* Acute thrombophlebitis
* History of pulmonary edema or decompensated congestive heart failure
* Currently has an active infection of the skin such as cellulitis requiring antibiotics
* Poorly controlled diabetes with an HbA1c value of >10%
* Exhibits any condition which, according to the PI, justifies the subjects exclusion from the study, such as a medical condition where an increase in venous or lymphatic return is undesirable.
* Subjects with open ulcers must be able to follow their care regimen for ulcer healing concurrently with the assigned study regimen.
* Participating in another clinical trial
* Changes to medications that affect edema within the last 30 days
* Currently pregnant or trying to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fedor Lurie, MD, PhD, Principal Investigator — Associate Director, Jobst Vascular Institute
Locations (11):
- United States (11):
  - Associated Foot and Ankle Specialists, LLC, Phoenix, Arizona
  - Empire Orthopedic Center, Colton, California
  - University of California, San Diego, La Jolla, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Long Beach VA Healthcare System, Long Beach, California
  - Park Nicollet Heart and Vascular Center, Minneapolis, Minnesota
  - Stony Brook Vein Center, Stony Brook, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio Health System, Columbus, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Greenville Hospital System, Greenville, South Carolina

REFERENCES:
- [Derived] Lurie F, Schwartz M. Patient-centered outcomes of a dual action pneumatic compression device in comparison to compression stockings for patients with chronic venous disease. J Vasc Surg Venous Lymphat Disord. 2017 Sep;5(5):699-706.e1. doi: 10.1016/j.jvsv.2017.06.003. PMID 28818225

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACTitouch | Standard Compression Garments
Started | 41 | 40
Completed | 32 | 34
Not Completed | 9 | 6
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants with bilateral disease received both treatment. The participate was randomly assigned a treatment to the right leg and were instructed to wear the other treatment on their left leg.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACTitouch | Standard Compression Garments | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.5) | 61.1 (11.7) | 62.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  United States | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Ease of Use and Comfort for Subjects Using the ACTitouch System.
Description: Ease of application and removal (donning and doffing) the treatment at the baseline visit. Comfort of treatment after the treatment was first applied.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: Percent of participants
Units Other Than Participants: Lower Extremities Analyzed
Arm/Group | ACTitouch | Standard Compression Garments
Number analyzed (Participants) | 41 | 40
Number analyzed (Lower Extremities Analyzed) | 66 | 70
Percent of participants
  % Reported Easy/Very Easy Donning - Baseline | 70.8 [58.8 to 80.4] | 37.5 [26.7 to 49.7]
  % Reported Easy/Very EasyDoffing - Baseline | 89.2 [79.4 to 94.7] | 59.4 [47.1 to 70.5]
  % Reported Comfortable/Very 1st Applied - Baseline | 70.8 [58.8 to 80.4] | 57.8 [45.6 to 69.1]
  % Reported Easy/Very Easy Donning - 30 Days | 64.9 [51.9 to 76.0] | 54.8 [42.5 to 66.6]
  % Reported Easy/Very Easy Doffing - 30 Day | 89.5 [78.9 to 95.1] | 66.1 [53.7 to 76.7]
  % Reported Comfortable/Very 1st Applied - 30 Days | 54.4 [41.6 to 66.6] | 63.9 [51.4 to 74.8]
  % Reported Comfortable/Very IPC 30 days | 62.3 [48.8 to 74.1] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | ACTitouch | Standard Compression Garments
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 5/41 | 0/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTitouch (N=41) | Standard Compression Garments (N=40)
Ulcer / Blister (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Participants could have either unilateral or bilateral disease. Bilateral participants had treatment randomly assigned to the right leg. The left leg received the treatment not assigned to their right leg (i.e: right leg - Grp A: Left Leg - Grp B).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less